CLINICAL TRIAL: NCT02936713
Title: Exploratory Study Aiming at Assessing the Impact of Specific and Controlled Diets Combined With a Fermented Milk Product on Gas-related Symptoms and Associated Measurements in FGID and Non-FGID Subjects
Brief Title: Effect of Controlled Diet Combined With a Fermented Milk Product on Gas-related Symptoms
Acronym: FLATBACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NU362
Record Dates: First submitted 2015-06-12; First posted 2016-10-18 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Functional Gastrointestinal Disorders
Keywords: flatulence; gas; probiotics; fermented milk; diet; functional gastrointestinal disorders
MeSH Terms: conditions — Gastrointestinal Diseases; Flatulence; Mucopolysaccharidosis IV | interventions — Cultured Milk Products; Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1=Functional Gastro-Intestinal Disorder (FGID) (Experimental): 1=FGID study group: 40 evaluable FGID subjects with a functional gastrointestinal disorder (FGID) complaining of excessive gas evacuation per anus (i.e excessive flatulence), aged from 18 to 75 years that will consume a 3-day specific and controlled mild flatulogenic diet twice at 25 days of interval (combined or not with a fermented milk product)
  Interventions: Other: Fermented milk product with probiotics (FMPP)
- 2=Non-FGID (Experimental): 2=Non-FGID study group: 60 evaluable non-FGID subjects aged from 18 to 75 years that will consume a 3-day specific controlled high flatulogenic diet twice at 25 days of interval (combined or not with a fermented milk product)
  Interventions: Other: Fermented milk product with probiotics (FMPP)

INTERVENTIONS:
Other: Fermented milk product with probiotics (FMPP) — 2 pots of 125g FMPP / day

SUMMARY:
To select among different dietary and clinical conditions the most appropriate to assess the impact of a fermented milk product on gas-related symptoms

DETAILED DESCRIPTION:
To select among different dietary (mild or high flatulogenic diet) and clinical conditions (FGID or non-FGID population) as well as different measured parameters (self-completed questionnaires assessing gas related symptoms, digestive well-being and bowel functions, gas volume distribution in the colon by MRI, volume and composition of gas collected per anus and frequency of gas evacuations per anus), the most appropriate to assess the impact of a fermented milk product on gas-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* 1=FGID group: Subject with body mass index (BMI) between 18.5 and 30.0 kg/m2 (bounds excluded); Subject with a functional gastrointestinal disorder according to ROME III criteria; Subject complaining of excessive intestinal gas evacuation (i.e. flatulence); Subject willing to follow strict dietary instructions; Subject who normally consumes dairy products;
* 2=Non-FGID group: Subject with body mass index (BMI) between 18.5 and 30.0 kg/m2 (bounds excluded); Subject with no functional gastrointestinal disorder according to ROME III criteria; Subject with no gastrointestinal disorders according to investigator's medical assessment; Subject willing to follow strict dietary instructions; Subject who normally consumes dairy products

Exclusion Criteria:

* 1=FGID group: Subject with any disease/disorder which can interfere with the gas collection; Subject with any antecedents of digestive surgery; Subject with any intake of antibiotics in the previous 2 months; Subject with any current use of any medication with potential central nervous system effects (except for chronic treatment with anxiolytics and antidepressants started at least 3 months before inclusion in the study); Subject taking drugs that might modify gastrointestinal function (except for chronic treatment with laxatives, started at least 3 months before inclusion in the study) ;
* 2=Non-FGID group: Subject with any disease/disorder which can interfere with the gas collection; Subject with any antecedents of digestive surgery; Subject with any intake of antibiotics in the previous 2 months; Subject with any current use of any medication with potential central nervous system effects; Subject taking drugs that might modify gastrointestinal function

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

PRIMARY OUTCOMES:
Change in number of gas evacuations per anus | during a 3-day baseline period and during two 3-day periods of controlled diet before and after a 28-day study product consumption period
  Change in number of gas evacuations per anus: number of events will be recorded daily using a gas event counter, during a 3-day baseline period and during two 3-day periods of controlled diet before and after a 28-day study product consumption period.
Change in intestinal gas volume | following a 3-day period of controlled diet before and after a 28- day study product consumption period
  Change in intestinal gas volume: gas volume evacuated per anus will be continuously collected and measured every 15 minutes during 4 hours by a specific device, at the time of a standardized breakfast and following a 3-day period of controlled diet before and after a 28- day study product consumption period.
Change in intestinal gas composition | following a 3- day period of controlled diet before and after a 28-day study product consumption period
  Change in intestinal gas composition: amount of different types of gas (H2, CO2, CH4, O2, N2, H2S, mercaptans) from the 4-hours intestinal gas collection sample will be determined by gas chromatography following a 3- day period of controlled diet before and after a 28-day study product consumption period.
Change in colonic gas volume/segmental distribution | following a 3-day period of controlled diet before and after a 28-day study product consumption period
  Change in colonic gas volume/segmental distribution: total gas volume and distribution in the different regions of the colon (ascending, transverse, descending, sigmoid/rectum) will be determined using intestinal MRI following a 3-day period of controlled diet before and after a 28-day study product consumption period.
Gas related symptoms (self-completed questionnaire) | 3 days
Digestive well-being (self-completed questionnaire) | 3 days
Composition of gut microbiota (molecular biology methods) | 5 days
Bowel function (self-completed questionnaire; bristol stool scale) | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron - DIGESTIVE SYSTEM RESEARCH UNIT, Barcelona, Spain